CLINICAL TRIAL: NCT04920591
Title: Efficacy of Doll thErapy Compared With Standard Treatment in the Control of Behavioral and Psychologic Symptoms and CaRegIver Burden of dEmentia
Brief Title: Doll Therapy in Dementia
Acronym: DESCRIBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Patrizia D'Amelio, associated professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0098548
Record Dates: First submitted 2021-06-02; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Dementia
Keywords: behavioral and psychologic symptoms in dementia; hospital; doll therapy; non-pharmacological approach; nursing homes
MeSH Terms: conditions — Dementia; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- doll therapy (DT) (Experimental): doll therapy (emathy dolls)
  Interventions: Other: doll treatment
- Standard treatment (ST) (No Intervention): standard clinical practice

INTERVENTIONS:
Other: doll treatment — The doll used in the study is the "empathy doll"; these dolls are designed to obtain an optimal interaction with patients and to arouse empathy.
  Arms: doll therapy (DT)

SUMMARY:
Behavioral and psychologic symptoms in dementia (BPSD) are frequent and represent a burden for patients and caregivers, the use of a first line non-pharmacologic approach is highly recommended. DESCRIBE is a randomized controlled trial on the effect of doll therapy (DT) on BPSD in different clinical settings.

The investigators will enroll fifty-two nursing homes residents and 52 acute in-patients with dementia and BPSD. Subjects will be randomized to DT or standard treatment (ST), The investigators will measured agitation, delirium and caregiver burden with standard clinical scales at baseline and during treatment. Nursing home residents will be evaluated after 45 and 90 days of treatment, in-patients will be evaluated at baseline and at hospital discharge. In acute in-patients, a follow-up of 4 weeks after hospital discharge will be carried out in order to evaluate the effect of DT withdrawal.

Primary outcomes will be the reduction of BPSD and the reduction of professional caregiver burden Secondary outcome will be the reduction of delirium and of effect of family caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

* age ≥65 years;
* diagnosis of dementia moderate to severe Clinical Dementia Rating scale (CDR) ≥2;
* presence of agitation and/or aggressiveness;
* manual and visual abilities sufficient in order to interact with the doll.

Exclusion Criteria:

* age <65 years;
* refuse to participate;
* mild forms of dementia (CDR<2);
* contraindication for DT as experience of mournful or traumatic events related to parental experience;
* life expectancy lower than 3 months;
* negative interaction with the doll.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of behavioral and psychologic symptoms in dementia measured by Neuropsychiatric Inventory (NPI) scale and by the A.Di.Co scale | 10-45-90 days
  Change in NPI and A.Di.Co scales
Change in professional caregivers burden measured by the Greutzner scale | 10-45-90 days
  change in professional caregiver burden

SECONDARY OUTCOMES:
Incidence of delirium measured by the Confusion assessment Method (CAM) scale | 45 and 90 days
  change in delirium incidence
Change in caregiver burden measured by the caregiver Burden Inventory (CBI) | 28 days
  Change in CBI

CONTACTS AND LOCATIONS:
Locations (1):
- città della salute e della Scienza, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santagata F, Massaia M, D'Amelio P. The doll therapy as a first line treatment for behavioral and psychologic symptoms of dementia in nursing homes residents: a randomized, controlled study. BMC Geriatr. 2021 Oct 12;21(1):545. doi: 10.1186/s12877-021-02496-0. PMID 34641791